CLINICAL TRIAL: NCT01468948
Title: Dose Escalation Study of Oral Octanoic Acid in Patients With Essential Tremor
Brief Title: Octanoic Acid for Essential Tremor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120024; 12-N-0024
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-07-18

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Tremor; Octanol; Octanoic Acid
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — octanoic acid

INTERVENTIONS:
Drug: Octanoic Acid

SUMMARY:
Background:

- Essential tremor (ET) is a condition of out-of-control shaking. Several drugs are used to treat ET. However, they are often only partly helpful and can have side effects. Many people with ET get some relief from drinking alcohol. Octanol, a food additive similar to alcohol, can improve tremor in animals and is less likely to make people feel drunk. One form of octanol, called 1-octanol, has been shown to improve tremor in some people and had few side effects. 1-octanol is converted to octanoic acid, and research suggests that octanoic acid itself might suppress ET with no significant side effects such as drunkenness. Researchers want to see what dose of octanoic acid is most useful in reducing ET.

Objectives:

- To test different doses of octanoic acid to treat essential tremor.

Eligibility:

* Individuals at least 21 years of age who have ET that responds to treatment with alcohol.
* Participants must be able to stop taking certain ET medications during the study.

Design:

* This study requires three visits. Visit 1 is a screening visit that will take up to 5 hours. Visit 2 is a 2- to 3-day inpatient admission to the National Institutes of Health Clinical Center. Visit 3 is a followup outpatient visit 1 to 2 weeks after the hospital admission.
* At the screening visit, participants will have a physical exam, neurological exam, and medical history. Blood and urine samples will be collected. Participants will also have an alcohol dose test to measure the tremor s response to alcohol.
* For the study visit, participants will enter the hospital for testing. Participants will have the study drug and test the tremor's response to it. Frequent blood samples will be collected.
* One to two weeks after leaving the hospital, participants will have a final followup study visit. Blood samples will be collected.

DETAILED DESCRIPTION:
OBJECTIVE:

To determine the maximum tolerated dose of oral octanoic acid (OA) in patients with essential tremor. Further study objectives include the evaluation of the efficacy and tolerability of octanoic acid with escalation doses, as well as the pharmacokinetic and pharmacodynamic profile.

STUDY POPULATION:

Up to 30 subjects with ethanol-responsive essential tremor (ET) will be included in the study. Subjects will be recruited in groups of 6 per dose level.

DESIGN:

The study objectives will be tested using a 3+3 dose escalation design. Per dose level, 3 subjects will be recruited, and dose levels will be 8, 16, 32, 64, and 128 mg/kg, with additional 3 subjects at the same level if one of the three subjects exhibits dose limit toxicity. Subjects will undergo a screening visit, followed by a 2 to 3-day inpatient admission during which the study drug OA will be administered. An outpatient follow-up visit will conclude the study.

OUTCOME MEASURES:

The primary outcome will be measured by evaluating dose-limiting toxicity, which will be reached once 2 or more subjects exhibit a grade 2 adverse event (CTCAE) on the same dose-level, which is related to OA. The dose below the level at which 2 or more grade 2 OA-related adverse events have been observed, will then be defined as maximum tolerated dose (MTD) and the study stopped. Toxicity for the primary outcome will be monitored by an unblinded independent data safety monitoring board (DSMB), who will determine when the primary outcome is reached.

Secondary measures will include safety measures such as routine laboratory parameters, EKG measures, vital signs as well as a standardized assessment for signs of intoxication. Additional secondary outcome measures will include efficacy measures such as tremor accelerometry and digital spiral analysis, as well as a standardized clinical tremor rating scale. Furthermore, pharmacokinetic sampling will be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of essential tremor with bilateral hand tremor as the predominant feature, which is known to be responsive to ethanol.
* Unequivocal accelerometric tremor of both hands on screening examination (bilateral central tremor component during postural tremor accelerometry, consistent with ET)
* Reduction of accelerometric tremor power of at least 35% following a formal ethanol challenge during the screening visit.
* Subjects must be willing and safely able to abstain from any medication for the treatment of tremor for a period of at least 5 plasma half-lives of the individual drug prior to study participation. (For Propranolol/Inderal , Gabapentin/Neurontin this will be 1 day; for Primidone/Mysoline : 26 days).

Subjects must be willing to refrain from alcohol and drinks or food containing caffeine starting 48 hours prior to the study visits

EXCLUSION CRITERIA:

* Patients with any other significant pathological finding in the neurological examination other than typical symptoms of ET
* Acute or chronic severe medical conditions which would preclude the subject from participating (e.g., severe heart disease NYHA grade 3 or 4, renal failure, hepatic failure, lung disease, uncontrolled hyperthyroidism)
* Subjects with concomitant therapy with warfarin or NSAIDs (other than aspirin), when taken on a regular basis and cannot be discontinued at least 14 days prior to study participation, because of potential interactions with octanoic acid (displacement of albumin binding in human serum)(Noctor et al. 1992)
* Established diagnosis of diabetes mellitus, as fasting-periods of up to 12 hours are required in the protocol.
* Subjects with active or past alcohol abuse or dependence (AUDIT score greater than or equal to 8)
* Elevated liver function parameters (AST, ALT, GGT), higher than the 1.5 fold upper limit of the normal range (as defined by the NIH Clinical Center Laboratory Medicine Department), or any other clinically significant abnormalities on their baseline laboratory tests. The limit for AST therefore will be 51 U/l, for ALT 62 U/L, and GGT 128 U/l.
* Female subjects who are pregnant or breastfeeding
* Subjects aged < 21 years
* Known flushing symptoms after alcohol intake or allergy to alcohol (any yes answer in the standardized Alcohol Flushing Questionnaire)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10-28; Primary Completion 2012-07-18 (Actual); Study Completion 2012-07-18 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 2 years

SECONDARY OUTCOMES:
Effect on tremor | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bain P, Brin M, Deuschl G, Elble R, Jankovic J, Findley L, Koller WC, Pahwa R. Criteria for the diagnosis of essential tremor. Neurology. 2000;54(11 Suppl 4):S7. No abstract available. PMID 10854345
- [Background] Ashitani J, Matsumoto N, Nakazato M. Effect of octanoic acid-rich formula on plasma ghrelin levels in cachectic patients with chronic respiratory disease. Nutr J. 2009 Jun 16;8:25. doi: 10.1186/1475-2891-8-25. PMID 19527531
- [Background] Bach AC, Babayan VK. Medium-chain triglycerides: an update. Am J Clin Nutr. 1982 Nov;36(5):950-62. doi: 10.1093/ajcn/36.5.950. PMID 6814231
- [Derived] Voller B, Lines E, McCrossin G, Tinaz S, Lungu C, Grimes G, Starling J, Potti G, Buchwald P, Haubenberger D, Hallett M. Dose-escalation study of octanoic acid in patients with essential tremor. J Clin Invest. 2016 Apr 1;126(4):1451-7. doi: 10.1172/JCI83621. Epub 2016 Feb 29. PMID 26927672